CLINICAL TRIAL: NCT06361823
Title: An Exploratory Study Assessing the Efficacy and Safety of Semaglutide for Idiopathic Intracranial Hypertension Treatment
Brief Title: Exploratory Study on the Efficacy and Safety of Semaglutide for Idiopathic Intracranial Hypertension Treatment
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Principal Investigator, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIH-Semaglutide
Record Dates: First submitted 2024-03-02; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Idiopathic Intracranial Hypertension
MeSH Terms: conditions — Pseudotumor Cerebri | interventions — semaglutide; Caloric Restriction

STUDY DESIGN:
Intervention Model Description: The researchers are tasked with adhering to the protocol requirements when selecting participants, and consistently enrolling eligible patients who are then randomly assigned to either the experimental or control group in a 1:1 ratio. The randomization process is overseen by expert statisticians and executed by specialized clinical researchers in an independent manner.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide (Experimental): Expanding on the usual treatment regimen, Semaglutide is administered through a subcutaneous injection once weekly over a period of 3 months. Initially, the dose is 0.25 mg for the first month, then increased to 0.5 mg for patients who could tolerate it in the second month, and finally raised to 1.0 mg for patients who still tolerated it in the third month.
  Interventions: Drug: Semaglutide; Dietary Supplement: Low calorie diet
- Usual treatment (Active Comparator): Usual treatment refers to the 2018 consensus guidelines on the management of IIH.
  Interventions: Dietary Supplement: Low calorie diet

INTERVENTIONS:
Drug: Semaglutide — Giving Semaglutide via subcutaneous injections on a weekly basis for a duration of 3 months. The dosage is 0.25 mg for the initial month, then upped to 0.5 mg for patients who could handle it in the second month, and eventually escalated to 1.0 mg for patients who continued to tolerate it in the third month.
  Other Names: Ozempic
  Arms: Semaglutide
Dietary Supplement: Low calorie diet — Low calorie diet (max 1200 kcal/day)

SUMMARY:
This study aims to investigate the safety and efficacy of semaglutide in patients with Idiopathic intracranial hypertension.

DETAILED DESCRIPTION:
Idiopathic intracranial hypertension (IIH) is a condition characterized by elevated pressure within the skull for reasons that are not yet understood. This condition does not involve abnormalities in the cerebrospinal fluid or any structural brain damage. Individuals with this condition commonly experience persistent headaches, and some may face the potential of irreversible vision loss, significantly impacting their psychological well-being and overall quality of life. At present, the efficacy of medications like acetazolamide and topiramate in managing IIH is constrained by practical clinical constraints. Recent studies have indicated that glucagon-like peptide-1 receptor agonists show promise as a potential treatment option for IIH. Semaglutide, as a long-acting glucagon-like peptide-1 formulation, has a half-life of up to 160 hours and only needs to be injected once a week. It is easy to administer and has good safety and tolerability. Hence, the objective of this study is to investigate the effectiveness and safety of semaglutide in managing idiopathic intracranial hypertension, laying the groundwork for subsequent extensive, multicenter research endeavors.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 18 to 75 years old, both male and female.
* Confirmed definite IIH with papilledema and lumbar opening pressure ≥25 cm cerebrospinal fluid according to Friedmann diagnostic criteria.
* Voluntarily sign a written informed consent form.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Currently using any hypoglycemic drugs, including glucagon like peptide-1 receptor agonists.
* Known to be allergic to the active ingredients or any excipients in Semaglutide.
* History or family history of Medullary Thyroid Carcinoma (MTC) or Multiple Endocrine Neoplasias (MEN1/MEN2).
* Diabetes, ketoacidosis, severe gastrointestinal diseases, pancreatitis, severe heart failure.
* Vision loss caused by other diseases, such as diabetes retinopathy, iritis, cataract, etc.
* Malignant IIH with vision at risk necessitating surgical intervention.
* Unable to cooperate in completing imaging examinations.
* History of bariatric surgery or cerebrospinal fluid diversion.
* Have used any drugs known to increase intracranial pressure within the past 3 months (including vitamin A, tetracycline drugs, lithium, etc).
* Have participated in other clinical trials within the past 3 months, or did not withdraw from other clinical trials at the time of signing the informed consent form.
* Other situations determined by the researcher that may pose a threat to the patients' life safety or may have an impact on the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Intracranial pressure | 12 weeks
  The intracranial pressure is represented by the cerebrospinal fluid pressure measured by lumbar puncture in a lateral position.
Adverse reactions | 12 weeks
  Adverse reactions include gastrointestinal reactions (such as nausea, vomiting, diarrhea), hypoglycemia, allergic reactions (such as rapid allergic reactions, vascular edema).

SECONDARY OUTCOMES:
Headache severity | Baseline + 12 weeks
  It is measured by the questionnaire "Headache Impact Test-6" (HIT-6); score range is 36-78. The higher the score, the more severe the headache.
Degree of papilledema | Baseline + 12 weeks
  It is represented by the Frisén Grade (0-5, 0 is the minimal, 5 is the worst) measured by fundoscope.
Perimetric mean deviation | Baseline + 12 weeks
  It is measured by Humphrey automated perimetry.
Optic nerve sheath diameter | Baseline + 12 weeks
  It is measured by optic nerve sheath ultrasound.
Body mass index | Baseline + 12 weeks
  Change in body mass index.

IPD SHARING:
Plan to Share IPD: No